CLINICAL TRIAL: NCT07255183
Title: Impact of Blood Glucose on Motivation States: A Double-Blind Placebo-Controlled Study
Brief Title: Glucose and Motivation States
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY009043
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Motivation
MeSH Terms: interventions — Exercise; Sugar-Sweetened Beverages

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise + sugar drink (Experimental)
  Interventions: Behavioral: Exercise; Dietary Supplement: Sugar Drink
- Exercise + non-sugar drink (Placebo Comparator)
  Interventions: Behavioral: Exercise; Dietary Supplement: Non-sugar beverage
- Rest + sugar drink (Active Comparator)
  Interventions: Dietary Supplement: Sugar Drink
- Rest + non-sugar drink (Placebo Comparator)
  Interventions: Dietary Supplement: Non-sugar beverage

INTERVENTIONS:
Behavioral: Exercise — Exercise 30 minutes at moderate intensity (10% below ventilatory threshold)
  Arms: Exercise + non-sugar drink; Exercise + sugar drink
Dietary Supplement: Sugar Drink — Consume 250mL beverage (water + 6 tablespoons table sugar)
  Arms: Exercise + sugar drink; Rest + sugar drink
Dietary Supplement: Non-sugar beverage — Consume 250mL beverage (water + 1.5 teaspoons of stevia powder)
  Arms: Exercise + non-sugar drink; Rest + non-sugar drink

SUMMARY:
The purpose of this study is to evaluate how motivation is impacted by exercise and beverage consumption. You will be asked to report to our lab for 5 visits each separated by 2+ days over a period of 2-3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18-30 m/kg^2
* Health Status: generally healthy; no cardiopulmonary/metabolic/orthopedic disease or limitations
* Blood Pressure: excluded with SBP of 130+ mmHg or DBP of 80+ mmHg
* Glucose Status: excluded and instructed to seek medical consultation if fasting values are <70 mg/dl or >125 mg/dl; included but encouraged to seek medical consultation if fasting values are 100-125 mg/dl

Exclusion Criteria:

* None

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
State Motivation to Move | 60 minutes
  Score on movement subscale of Cravings for Rest and Volitional Energy Expenditure Survey (0 is lowest, 100 is highest)

SECONDARY OUTCOMES:
State motivation to rest | 60 minutes
  Score on rest subscale of Cravings for Rest and Volitional Energy Expenditure Survey (0 is lowest, 100 is highest)

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data (including data dictionaries) will be shared. This includes individual participant data that underlie the results reported in any aspect of a published article (text, tables, figures, and appendices).
  Other documents that will be available include the study protocol, statistical analysis plan, informed consent form, and analytic code. The data will be available immediately after publication with no end date. Data will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed to Dr. Garrett Ash at Yale University (garrett.ash@yale.edu). To gain access, data requesters will need to sign a data access agreement.